CLINICAL TRIAL: NCT02735317
Title: Efficacy and Safety of FORRAD® for the Management of Radiation-induced Mucositis in Patients With Nasopharyngeal Carcinoma Receiving IMRT: A Single-center, Randomized Controlled Trial
Brief Title: Efficacy and Safety of FORRAD® for the Management of Radiation-induced Mucositis in Patients With Nasopharyngeal Carcinoma Receiving IMRT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yun-fei Xia (Other)
Responsible Party: Sponsor-Investigator, Yun-fei Xia, Director of the Department of Radiation Oncology, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2015-074-01
Record Dates: First submitted 2016-03-27; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Nasopharyngeal Neoplasms; Stomatitis
Keywords: Nasopharyngeal carcinoma (NPC); radiotherapy; oral mucositis (OM)
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Stomatitis; Nasopharyngeal Carcinoma | interventions — Gentamicins; Vitamin B 12; Procaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FORRAD group (Experimental): This group of patients will receive Oral Ulcer Gargle (FORRAD®) during study for prevention and treatment of acute radiation-induced oral mucositis (OM).
  This is the experimental group.
  Interventions: Drug: Oral Ulcer Gargle (FORRAD®)
- Quadruple mixture group (Active Comparator): This group of patients will receive quadruple mixture, which is composed of dexamethasone, gentamicin, vitamin B12, and procaine, during study for prevention and treatment of acute radiation-induced oral mucositis (OM).
  This is the active comparator group.
  Interventions: Drug: Quadruple mixture, composed of dexamethasone, gentamicin, vitamin B12, and procaine

INTERVENTIONS:
Drug: Oral Ulcer Gargle (FORRAD®) — Oral Ulcer Gargle (FORRAD®) is prescribed at the beginning of radiotherapy for free. Patients are asked to start application of Oral Ulcer Gargle (FORRAD®) at the onset of radiotherapy, four times a day (after meals and before bedtime), until completion of their radiotherapy. All patients will receive conventional health education and medical care for prevention and treatment of radiation-induced oral mucositis. When grade > 3 OM happened, other interventions, such as prophylactic or therapeutic antibacterial therapy, will be used, and radiotherapy should be interrupted.
  Arms: FORRAD group
Drug: Quadruple mixture, composed of dexamethasone, gentamicin, vitamin B12, and procaine — Quadruple mixture is prescribed at the beginning of radiotherapy. Patients are asked to start application of quadruple mixture at the onset of radiotherapy, four times a day (before meals and before bedtime), until completion of their radiotherapy. All patients will receive conventional health education and medical care for prevention and treatment of radiation-induced oral mucositis. When grade > 3 OM happened, other interventions, such as prophylactic or therapeutic antibacterial therapy, will be used, and radiotherapy should be interrupted.
  Arms: Quadruple mixture group

SUMMARY:
Radiation therapy remains the principal treatment for nasopharyngeal carcinoma (NPC). The most frequently occurred radiation-related side effect is probably the radiation-induced oral mucositis (OM), which affects up to 100% of NPC patients receiving radiation therapy. When severe, oral mucositis increases the risk of infection and may compromise clinical outcomes by necessitating treatment breaks, dosage reductions, and reduced therapy compliance. In China, a quadruple mixture, composed of dexamethasone, gentamicin, vitamin B12, and procaine, is commonly prescribed when NPC patients begin to suffer from radiation-induced OM. However, the incidence of radiation-induced OM is still quite high. Oral Ulcer Gargle (FORRAD®) is a proprietary viscous liquid mucoadhesive hydrogel formulation. It creates a palliative barrier over injured mucosa, to prevent and to cure radiation-induced OM. The objective of this randomized phase II study is to assess the efficacy and safety of Oral Ulcer Gargle (FORRAD®) as an intervention for radiation-induced OM in the treatment of NPC, compared with the commonly used quadruple mixture, which is composed of dexamethasone, gentamicin, vitamin B12, and procaine.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is one of the most common malignances in South China. Radiation therapy remains the principal treatment for NPC. The most frequently occurred radiation-related side effect is probably the radiation-induced oral mucositis (OM), which affects up to 100% of NPC patients receiving radiation therapy. Although intensity modulated radiation therapy (IMRT) has been widely used in China nowadays, the incidence of radiation-induced oral mucositis is still high. OM can decrease patients' oral intake and nutrition, leading to dehydration, weight loss, and declining performance status that may require intravenous fluid hydration, feeding tube placement, and hospitalization. OM also may increase opioid use. When severe, oral mucositis increases the risk of infection and may compromise clinical outcomes by necessitating treatment breaks, dosage reductions, and reduced therapy compliance. Common clinical management strategies include bland rinses, topical anesthetics and analgesics, mucosal coating agents, and systemic analgesics. However, none of these interventions has been supported by conclusive evidence. In China, a quadruple mixture, composed of dexamethasone, gentamicin, vitamin B12, and procaine, is commonly prescribed when NPC patients begin to suffer from radiation-induced OM.

Oral Ulcer Gargle (FORRAD®) is a proprietary viscous liquid mucoadhesive hydrogel formulation. It creates a palliative barrier over injured mucosa, to prevent and to cure radiation-induced OM.

The objective of this randomized phase II study is to assess the efficacy and safety of Oral Ulcer Gargle (FORRAD®) as an intervention for radiation-induced OM in the treatment of NPC, compared with the commonly used quadruple mixture, which is composed of dexamethasone, gentamicin, vitamin B12, and procaine.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed and previously untreated nasopharyngeal carcinoma.
2. Age ≥ 18 years and ≤ 65 years.
3. Karnofsky performance status (KPS) score ≥ 70.
4. Planned to receive radiotherapy alone or concurrent chemoradiotherapy, with intensity-modulated radiation therapy (IMRT).
5. Adequate bone marrow function: while blood cell >= 3,000/μL, absolute neutrophil count >= 1,500/μL, hemoglobin >= 100g/L, platelet >= 75,000/μL.
6. Life expectancy of >= 3 months.

Exclusion Criteria:

1. Known allergic reaction to any component of Oral Ulcer Gargle (FORRAD®) or quadruple mixture, which is composed of dexamethasone, gentamicin, vitamin B12, and procaine, or severe allergic constitution.
2. Other conditions that the investigators consider as inappropriate for enrolling into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade ≥ 3 mucositis | Day 56 after completion or termination of radiotherapy
  Incidence of grade ≥ 3 mucositis according to CTCAE version 4.0
OMAS | Day 56 after completion or termination of radiotherapy
  Oral Mucositis Assessment Scale (OMAS) provides an objective assessment of oral mucositis based on assessment of the appearance and extent of redness and ulceration in various areas of the mouth.
OMDQ MTS question 2 (Q2) score | Day 56 after completion or termination of radiotherapy
  Oral Mucositis Daily Questionnaire (OMDQ) mouth and throat soreness (MTS) question 2 (Q2) is a 5-point categorical scale in which patients grade MTS from 0 (no soreness) to 4 (extreme soreness)3 which is a component of the OMDQ in that it tracks very well with objective (WHO score and opioid use) and subjective measurement of OM severity.
WHO score | Day 56 after completion or termination of radiotherapy
  The World Health Organization (WHO) Oral Toxicity score combines both elements into a single score that grades the severity of the condition from 0 (no oral mucositis) to 4 (swallowing not possible such that patient needs supplementary nutrition).
EORTC QLQ-C30 | Day 56 after completion or termination of radiotherapy
  EORTC QLQ-C30 is a Quality-of-Life Instrument proposed by the European Organization for Research and Treatment of Cancer (EORTC), for use in International Clinical Trials in Oncology. The QLQ-C30 incorporates nine multi-item scales: five functional scales (physical, role, cognitive, emotional, and social); three symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale.

SECONDARY OUTCOMES:
Interruption time during the schedule of radiotherapy | Through radiotherapy completion or termination, an average of 7 weeks
  The cumulative interruption time during the schedule of radiotherapy because of grade 4 or higher radiation-induced oral mucositis.
Time for healing of radiation-induced oral mucositis | Through study completion, an average of 15 weeks
  Time until healing of radiation-induced oral mucositis, after the completion or the termination of radiotherapy.
The cumulative dose of opioid used | Through study completion, an average of 15 weeks
  The cumulative dose of opioid used from the beginning of radiotherapy until the completion of study.
The cumulative time using opioid | Through study completion, an average of 15 weeks
  The cumulative time using opioid from the beginning of radiotherapy until the completion of study.
The change of body weight from baseline. | Baseline and 7 weeks
  The change of body weight before radiotherapy and the day when radiotherapy is completed or terminated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Zhang LF, Li YH, Xie SH, Ling W, Chen SH, Liu Q, Huang QH, Cao SM. Incidence trend of nasopharyngeal carcinoma from 1987 to 2011 in Sihui County, Guangdong Province, South China: an age-period-cohort analysis. Chin J Cancer. 2015 May 14;34(8):350-7. doi: 10.1186/s40880-015-0018-6. PMID 26058679
- [Background] Blanchard P, Lee A, Marguet S, Leclercq J, Ng WT, Ma J, Chan AT, Huang PY, Benhamou E, Zhu G, Chua DT, Chen Y, Mai HQ, Kwong DL, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Zhang L, Hui EP, Lu TX, Bourhis J, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy and radiotherapy in nasopharyngeal carcinoma: an update of the MAC-NPC meta-analysis. Lancet Oncol. 2015 Jun;16(6):645-55. doi: 10.1016/S1470-2045(15)70126-9. Epub 2015 May 6. PMID 25957714
- [Background] Mao YP, Yin WJ, Guo R, Zhang GS, Fang JL, Chi F, Qi ZY, Liu MZ, Ma J, Sun Y. Dosimetric benefit to organs at risk following margin reductions in nasopharyngeal carcinoma treated with intensity-modulated radiation therapy. Chin J Cancer. 2015 May 20;34(5):189-97. doi: 10.1186/s40880-015-0016-8. PMID 26058563
- [Background] Zheng Y, Han F, Xiao W, Xiang Y, Lu L, Deng X, Cui N, Zhao C. Analysis of late toxicity in nasopharyngeal carcinoma patients treated with intensity modulated radiation therapy. Radiat Oncol. 2015 Jan 13;10:17. doi: 10.1186/s13014-014-0326-z. PMID 25582731
- [Background] Porock D. Factors influencing the severity of radiation skin and oral mucosal reactions: development of a conceptual framework. Eur J Cancer Care (Engl). 2002 Mar;11(1):33-43. PMID 11966833
- [Background] Rodriguez-Caballero A, Torres-Lagares D, Robles-Garcia M, Pachon-Ibanez J, Gonzalez-Padilla D, Gutierrez-Perez JL. Cancer treatment-induced oral mucositis: a critical review. Int J Oral Maxillofac Surg. 2012 Feb;41(2):225-38. doi: 10.1016/j.ijom.2011.10.011. Epub 2011 Nov 8. PMID 22071451
- [Background] Wu F, Wang R, Lu H, Wei B, Feng G, Li G, Liu M, Yan H, Zhu J, Zhang Y, Hu K. Concurrent chemoradiotherapy in locoregionally advanced nasopharyngeal carcinoma: treatment outcomes of a prospective, multicentric clinical study. Radiother Oncol. 2014 Jul;112(1):106-11. doi: 10.1016/j.radonc.2014.05.005. Epub 2014 Jun 2. PMID 24933452
- [Background] Guo R, Tang LL, Mao YP, Zhou GQ, Qi ZY, Liu LZ, Lin AH, Liu MZ, Ma J, Sun Y. Clinical Outcomes of Volume-Modulated Arc Therapy in 205 Patients with Nasopharyngeal Carcinoma: An Analysis of Survival and Treatment Toxicities. PLoS One. 2015 Jul 6;10(7):e0129679. doi: 10.1371/journal.pone.0129679. eCollection 2015. PMID 26146828
- [Background] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Concurrent chemoradiotherapy plus adjuvant chemotherapy versus concurrent chemoradiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma: a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2012 Feb;13(2):163-71. doi: 10.1016/S1470-2045(11)70320-5. Epub 2011 Dec 7. PMID 22154591
- [Background] Allison RR, Ambrad AA, Arshoun Y, Carmel RJ, Ciuba DF, Feldman E, Finkelstein SE, Gandhavadi R, Heron DE, Lane SC, Longo JM, Meakin C, Papadopoulos D, Pruitt DE, Steinbrenner LM, Taylor MA, Wisbeck WM, Yuh GE, Nowotnik DP, Sonis ST. Multi-institutional, randomized, double-blind, placebo-controlled trial to assess the efficacy of a mucoadhesive hydrogel (MuGard) in mitigating oral mucositis symptoms in patients being treated with chemoradiation therapy for cancers of the head and neck. Cancer. 2014 May 1;120(9):1433-40. doi: 10.1002/cncr.28553. PMID 24877167